CLINICAL TRIAL: NCT02168946
Title: A Phase 3, Multi-Center, Randomized, Open-Label Study of Vabomere(Meropenem-vaborbactam) Versus Best Available Therapy in Subjects With Selected Serious Infections Due to Carbapenem-Resistant Enterobacteriaceae (CRE)
Brief Title: Efficacy, Safety, Tolerability of Vabomere Compared to Best Available Therapy in Treating Serious Infections in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rempex (a wholly owned subsidiary of Melinta Therapeutics, Inc.) (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Melinta Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rempex 506
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Urinary Tract Infection Complicated; Acute Pyelonephritis; Hospital Acquired Bacterial Pneumonia; Ventilator-associated Bacterial Pneumonia; Bacteremia; Abdominal Infection
MeSH Terms: conditions — Bacteremia; Intraabdominal Infections | interventions — meropenem and vaborbactam; vaborbactam; beta-Lactamase Inhibitors; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded adjudication committee
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vabomere (Experimental): Vabomere (meropenem 2g plus vaborbactam 2g) IV q8h, for up to 14 days
  Interventions: Drug: Vabomere
- Best Available Therapy (Active Comparator): Subjects will receive Best Available Therapy (IV antibiotics)
  Interventions: Drug: Best Available Therapy

INTERVENTIONS:
Drug: Vabomere — Vabomere for IV injection, administered as a 2 g/2 g dose
  Other Names: Combination meropenem and vaborbactam; beta-lactamase inhibitor and carbapenem antibiotic
  Arms: Vabomere
Drug: Best Available Therapy — Antibiotic(s) chosen by Investigator
  Other Names: IV Antibiotics
  Arms: Best Available Therapy

SUMMARY:
Vabomere™, (meropenem-vaborbactam) is being compared to the Best Available Therapy in the treatment of adults with selected serious infections due to Carbapenem Resistant Enterobacteriaceae

DETAILED DESCRIPTION:
In the current era of increased resistance to extended spectrum cephalosporins and penicillin/beta-lactamase inhibitor combinations, carbapenem antimicrobial agents are frequently the antibiotics of "last defense" for the most resistant pathogens in serious infections. However, the recent dissemination of serine carbapenemases (e.g. KPC) in Enterobacteriaceae within many hospitals worldwide now poses a considerable threat to carbapenems and other members of the beta-lactam class of antimicrobial agents.

Infections caused by Carbapenem-Resistant Enterobacteriaceae (CRE) are associated with high mortality rates and have limited treatment options. The loss of the carbapenem class of antimicrobial agents for treatment of Enterobacteriaceae (the most frequently occurring pathogens in the hospital setting), Acinetobacter baumannii, and Pseudomonas aeruginosa represents a critical setback in modern patient care.

As a result of the current lack of an optimal treatment for patients who have infections due to a CRE, physicians manage these patients with the limited anti-infective options available, including aminoglycosides, polymyxin B, colistin, tigecycline, or various combinations of these. There are limited efficacy data available for many of these therapies when used to treat serious CRE infections, particularly in combination, but with limited or no alternative therapies currently available, such treatments have become the Best Available Therapy despite the toxicities associated with many of them.

Vaborbactam is a novel beta-lactamase inhibitor that has inhibitory activity against many serine beta-lactamases and was optimized for inhibition of the KPC beta-lactamase and the potentiation of carbapenems against Enterobacteriaceae. Vaborbactam is being developed for use with meropenem (a broad spectrum injectable carbapenem antibiotic) to address the challenges of treatment of serious infections caused by pathogens increasingly resistant to available treatments.

Vabomere, (meropenem-vaborbactam) administered as a fixed combination by intravenous (IV) infusion, is being developed to treat serious gram-negative infections, such as complicated urinary tract infections (cUTI), acute pyelonephritis (AP), hospital-acquired bacterial pneumonia (HABP), ventilator-associated bacterial pneumonia (VABP), and bacteremia, including those infections caused by bacteria resistant to currently available carbapenems.

ELIGIBILITY:
* Inclusion Criteria:

  1. Willingness to comply with all study activities and procedures and to provide signed, written informed consent prior to any study procedures. If a subject is unable to provide informed consent due to their medical condition, the subject's legal representative will be provided with study information in order for consent to be obtained.
  2. Hospitalized male or female, ≥18 years of age.
  3. Weight ≤185 kg.
  4. Have a confirmed diagnosis of a serious infection, specifically cUTI or AP, cIAI, HABP, VABP, and/or bacteremia, requiring administration of IV antibacterial therapy.
  5. Have a known or suspected Carbapenem-Resistant Enterobacteriaceae (CRE) infection.
  6. Expectation, in the opinion of the Investigator, that the subject's infection will require treatment with IV antibiotics for a minimum of 7 days.
  7. Expectation that subjects with an estimated creatinine clearance <10 ml/min (Cockcroft-Gault) will receive hemodialysis at least 2 times per week.
  8. For cUTI & AP subjects only: expectation, in the judgment of the Investigator, that any indwelling urinary catheter or instrumentation (including nephrostomy tubes and/or indwelling stents) will be removed or replaced (if removal is not clinically acceptable) before or as soon as possible, but not longer than 12 hours, after randomization.

     For cIAI subjects only: • Expectation, in the judgment of the investigator, that operative drainage/debridement/removal (including open laparotomy, percutaneous drainage, or laparoscopic surgery) of any intra-abdominal collection or other potential source of intra abdominal infection will be performed;

     • Expectation that cultures from the aforementioned procedure (including open laparotomy, percutaneous drainage, or laparoscopic surgery) will be sent for microbiological evaluation, including gram stain, culture and susceptibility testing, and Vabomere susceptibility testing.
  9. Female subjects of childbearing potential, including those who are less than 2 years post menopausal, must agree to, and comply with, using 2 highly effective methods of birth control (i.e., condom plus spermicide, combined oral contraceptive, implant, injectable, indwelling intrauterine device, sexual abstinence, or a vasectomized partner) while participating in this study. In addition, all women of childbearing potential must agree to continue to use 2 forms of birth control throughout the study and for at least 30 days after administration of the last dose of study drug.
* Exclusion Criteria:

  1. History of any significant hypersensitivity or severe allergic reaction to any beta-lactam antibiotics (e.g., cephalosporins, penicillins, carbapenems, or monobactams).
  2. Known or suspected likely infection with New Delhi metallo- (NDM), Verona integron-encoded metallo- (VIM), or IMP-metallo-beta-lactamases or oxacillinase- (OXA)-beta-lactamases (i.e., Class B or Class D beta-lactamases).
  3. For subjects to be enrolled with the primary indication of cUTI or AP, any of the following urologic conditions:

     1. Likely to receive ongoing antibacterial drug prophylaxis after treatment of cUTI (e.g., subjects with vesico-ureteral reflux);
     2. Suspected or confirmed prostatitis;
     3. Requirement for bladder irrigation with antibiotics or for antibiotics to be administered directly via urinary catheter;
     4. Previous or planned cystectomy or ileal loop surgery;
     5. Uncomplicated urinary tract infection (for example, female subjects with urinary frequency, urgency or pain or discomfort without systemic symptoms or signs of infection);
     6. Complete, permanent obstruction of the urinary tract;
     7. Suspected or confirmed perinephric or renal corticomedullary abscess;
     8. Polycystic kidney disease; or
     9. Any recent history of trauma to the pelvis or urinary tract.
  4. For subjects to be enrolled with the primary indication of cIAI, any of the following conditions:

     1. Incomplete drainage of suspected or known intra-abdominal source;
     2. Likely to receive ongoing antibacterial drug prophylaxis or chronic suppressive therapy after intravenous treatment of cIAI;
     3. Source of infection thought to be related to or involving a non-removable prosthesis (e.g. intra-abdominal mesh) or implantable device, line (e.g. peritoneal catheter) or stent (e.g. biliary stent);
     4. Uncomplicated intra-abdominal infection, such as simple appendicitis, simple cholecystitis or gangrenous cholecystitis without rupture;
     5. Patients with infected necrotizing pancreatitis or pancreatic abscess;
     6. Patients whose surgery will include staged abdominal repair or "open abdomen" technique, or marsupialization (i.e. patients who undergo a surgical procedure where fascial closure is performed are eligible. The skin incision may be left open for purposes of wound management as long as fascial closure is accomplished);
     7. Patients in whom the intra-abdominal process is deemed not likely to be infectious in origin (e.g. bowel obstruction, ischemic bowel without perforation, traumatic bowel perforation within past 12 hours, perforated gastroduodenal ulcer within 24 hours); or
     8. Non-intra-abdominal infection (e.g. infection or abscess of the abdominal wall without extension into the intra-abdominal cavity).
  5. For subjects to be enrolled with the primary indication of HABP or VABP, any of the following conditions:

     1. Diagnosis of ventilator-associated tracheobronchitis
     2. Inability to obtain proper respiratory specimens for culture.
  6. For subjects to be enrolled with the indication of bacteremia unrelated to cUTI or AP, cIAI, HABP, and VABP, any of the following:

     1. Unverified CRE infection
     2. Source of infection thought to be related to or involving a non-removable or implantable device or line.
  7. Evidence of immediately life-threatening disease where in the opinion of the Investigator, the subject is unlikely to survive more than 72 hours from randomization.
  8. Acute Physiology and Chronic Health Evaluation (APACHE) II score >30.
  9. Known or suspected endocarditis, meningitis, intra-abdominal infection, or osteomyelitis.
  10. Irremovable or implantable device or line thought to be the potential source of infection.
  11. Evidence of significant hepatic, hematological, or immunologic disease or dysfunction.
  12. Women who are pregnant or breastfeeding.
  13. Require the use of inhaled antibiotics.
  14. Participation in any study involving administration of an investigational agent or device within 30 days prior to randomization into this study or previous participation in the current study.
  15. Previous participation in a study of vaborbactam.
  16. Any condition that, in the opinion of the Investigator, would compromise the safety of the subject or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-07; Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fusaro, Study Director — Sponsor GmbH; Keith Kaye, Principal Investigator — Wayne State University
Locations (44):
- United States (19):
  - Hartford, Connecticut
  - Tampa, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Evanston, Illinois
  - Indianapolis, Indiana
  - Detroit, Michigan
  - Royal Oak, Michigan
  - New Brunswick, New Jersey
  - Buffalo, New York
  - Flushing, New York
  - New York, New York
  - The Bronx, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charlottesville, Virginia
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - La Plata
  - Mendoza
- Brazil (5):
  - São José do Rio Preto, São Paulo
  - Belo Horizonte
  - Curitiba
  - Porto Alegre
  - São Paulo
- Colombia (3):
  - Barranquilla
  - Bogotá
  - Medellín
- Greece (2):
  - Athens
  - Thessaloniki
- Israel (4):
  - Haifa
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (6):
  - Bologna
  - Florence
  - Genova
  - Pisa
  - Rome
  - Udine
- Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhowmick T. Clinical Outcomes of Patient Subgroups in the TANGO II Study. Infect Dis Ther. 2021 Mar;10(1):35-46. doi: 10.1007/s40121-021-00405-x. Epub 2021 Feb 9. PMID 33565042
- [Derived] Wunderink RG, Giamarellos-Bourboulis EJ, Rahav G, Mathers AJ, Bassetti M, Vazquez J, Cornely OA, Solomkin J, Bhowmick T, Bishara J, Daikos GL, Felton T, Furst MJL, Kwak EJ, Menichetti F, Oren I, Alexander EL, Griffith D, Lomovskaya O, Loutit J, Zhang S, Dudley MN, Kaye KS. Effect and Safety of Meropenem-Vaborbactam versus Best-Available Therapy in Patients with Carbapenem-Resistant Enterobacteriaceae Infections: The TANGO II Randomized Clinical Trial. Infect Dis Ther. 2018 Dec;7(4):439-455. doi: 10.1007/s40121-018-0214-1. Epub 2018 Oct 1. PMID 30270406

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient enrolled November 2014 and last patient in June 2017. The patients were enrolled at 27 study sites in 8 countries. 77 patients (28 with bacteremia, 34 with cUTI, 8 with HABP/VABP and 7 with cIAI) were enrolled and 47 had confirmed Carbapenem-Resistant Enterobacteriaceae and therefore were included in the mCRE population.
Pre-assignment Details: Randomization was stratified by presenting indication (cUTI or AP, cIAI, HABP, VABP, or bacteremia) and by region (North America, Europe, Asia Pacific, and Rest of World).
Period: Overall Study
Arm/Group | Vabomere | Best Available Therapy
Started | 50 (2 additional subjects were randomized to Vabomere but did not receive study drug) | 25
Completed | 38 | 20
Not Completed | 12 | 5
Not completed — Adverse Event | 8 | 5
Not completed — Lost to Follow-up | 3 | 0
Not completed — Subject unable to come back for visits | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects who received at least one dose of study drug (MITT and Safety Population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Vabomere | Best Available Therapy | Total
Number analyzed (Participants) | 50 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 14 | 40
  >=65 years | 24 | 11 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (15.30) | 63.2 (13.10) | 63.5 (14.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 7 | 32
  Male | 25 | 18 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 41 | 20 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 43 | 22 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.90 (8.340) | 27.14 (7.522) | 27.64 (8.029)
Systemic Inflammatory Response Syndrome (SIRS) present [Count of Participants; unit: Participants] — SIRS is a serious condition related to systemic inflammation, organ dysfunction, and organ failure.
  Participants | 22 | 10 | 32
Creatinine Clearance <50 mL/min [Count of Participants; unit: Participants] | 12 | 9 | 21
Baseline Pathogen - Klebsiella pneumoniae [Count of Participants; unit: Participants] | 30 | 14 | 44

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects in the Microbiological Carbapenem-resistant Enterobacteriaceae Modified Intent-to-Treat (mCRE-MITT) Population With a Response of Overall Success [Complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP) Subjects]
Description: Overall success is defined as clinical cure & microbiological eradication. Eradication defined by FDA as the demonstration that the bacterial pathogen(s) found at baseline is reduced to <10x4 colony forming unit (CFU)/mL urine. Clinical cure defined as complete resolution or significant improvement of the baseline signs & symptoms, no further antimicrobial warranted.
Time Frame: at Test of Cure (TOC) visit (Day 12-23)
Population: The mCRE-MITT population includes all patients who had confirmed Carbapenem-Resistant Enterobacteriaceae at Baseline. (cUTI/AP patients only)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 12 | 4
Participants | 4 | 2

2. Primary Outcome: All-cause Mortality Rate in the mCRE-MITT Population [Hospital-acquired Bacterial Pneumonia (HABP), Ventilator-associated Bacterial Pneumonia (VABP) and Bacteremia Subjects)
Description: The All-cause mortality rate at Day 28 in the mCRE-MITT population (HABP/VABP and Bacteremia)
Time Frame: Day 28
Population: mCRE-MITT Population (HABP/VABP and Bacteremia subjects only)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 18 | 9
Participants | 4 | 4

3. Primary Outcome: Proportion of Subjects in the mCRE-MITT Population With a Clinical Outcome of Cure [Complicated Intra-abdominal Infection (cIAI) Subjects Only]
Description: Clinical cure defined as complete resolution or significant improvement of the baseline signs and symptoms, no further antimicrobial warranted.
Time Frame: at TOC visit (Day 12-23)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 2 | 2
Participants | 2 | 0

4. Secondary Outcome: The All-cause Mortality Rate in the mCRE-MITT Population (All Indications)
Description: All Cause Mortality at Day 28 in the mCRE-MITT population (all indications)
Time Frame: at Day 28
Population: mCRE-MITT population (all indications)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 32 | 15
Participants | 5 | 5

5. Secondary Outcome: The All-cause Mortality Rate in the m-MITT Population (All Indications)
Description: The All Cause Mortality rate at Day 28 in the m-MITT population (all indications)
Time Frame: at Day 28
Population: The m-MITT population includes all patients who receive at least one dose of study drug and have a baseline gram negative bacterial pathogen.
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 35 | 19
Participants | 5 | 5

6. Secondary Outcome: The All-cause Mortality Rate in the mCRE-MITT Population (cUTI/AP)
Description: All Cause Mortality at Day 28 in the mCRE-MITT population (cUTI/AP subjects only)
Time Frame: at Day 28
Population: mCRE-MITT (cUTI/AP subjects only)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 12 | 4
Participants | 1 | 0

7. Secondary Outcome: Proportion of Subjects in the mCRE-MITT Population With a Clinical Outcome of Cure (All Indications)
Description: Clinical cure defined as complete resolution or significant improvement of the baseline signs & symptoms, no further antimicrobial warranted.
Time Frame: at End of Therapy (EOT) visit (7-14 days) and TOC visit (12-23 days)
Population: mCRE-MITT population (all indications)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 32 | 15
Participants
  EOT | 21 | 5
  TOC | 19 | 4

8. Secondary Outcome: Proportion of Subjects in the mCRE-MITT Population With a Clinical Outcome of Cure (cUTI/AP Subjects Only)
Description: as for outcome 7
Time Frame: at EOT visit (7-14) and TOC visit (day 12-23)
Population: mCRE-MITT population (cUTI/AP subjects only)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 12 | 4
Participants
  EOT | 9 | 2
  TOC | 5 | 2

9. Secondary Outcome: Proportion of Subjects in the mCRE-MITT Population With a Clinical Outcome of Cure (HABP/VABP and Bacteremia)
Description: as for outcome 7
Time Frame: at EOT visit (7-14) and TOC visit (day 12-23)
Population: mCRE-MITT (HABP/VABP or Bacteremia Subjects only)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 18 | 9
Participants
  EOT | 10 | 3
  TOC | 12 | 2

10. Secondary Outcome: Proportion of Subjects in the Microbiological Modified Intent-to-Treat (m-MITT) Population With a Clinical Outcome of Cure (All Indications)
Description: as for outcome 3
Time Frame: at EOT visit (7-14) and TOC visit (day 12-23)
Population: m-MITT Population (all indications)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 35 | 19
Participants
  EOT | 24 | 7
  TOC | 21 | 6

11. Secondary Outcome: Proportion of Subjects in the m-MITT Population With a Clinical Outcome of Cure (cUTI/AP)
Description: as for outcome 7
Time Frame: at EOT visit (7-14) and TOC visit (day 12-23)
Population: m-MITT Population (cUTI/AP subjects only)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 13 | 8
Participants
  EOT | 10 | 4
  TOC | 6 | 4

12. Secondary Outcome: Proportion of Subjects in the m-MITT Population With a Clinical Outcome of Cure (HABP/VABP and Bacteremia)
Description: as for outcome 7
Time Frame: at EOT visit (7-14) and TOC visit (day 12-23)
Population: m-MITT Population (HABP/VABP or Bacteremia Subjects only)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 20 | 9
Participants
  EOT | 12 | 3
  TOC | 13 | 2

13. Secondary Outcome: Proportion of Subjects in the mCRE-MITT Population With a Microbiological Outcome of Eradication (All Indications)
Description: Includes subjects with microbiologic eradication or presumed eradication as defined: microbiologic eradication of the baseline pathogen or absence of culture result (microbiologic outcome of indeterminate or not assesses) where subject is deemed as clinical cure at that visit. For cUTI/AP subjects, demonstration that the bacterial pathogen(s) found at baseline is reduced to <10x4 CFU/mL urine (FDA).
Time Frame: at EOT visit (7-14) and TOC visit (day 12-23)
Population: mCRE-MITT Population (all indications)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 32 | 15
Participants
  EOT | 21 | 6
  TOC | 17 | 5

14. Secondary Outcome: Proportion of Subjects in the m-MITT Population With a Microbiological Outcome of Eradication (All Indications)
Description: Microbiological eradication defined for cUTI/AP as the demonstration that the bacterial pathogen(s) found at baseline is reduced to <10x4 CFU/mL urine (FDA).
Time Frame: at EOT visit (7-14) and TOC visit (day 12-23)
Population: m-MITT Population (all indications)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 35 | 19
Participants
  EOT | 23 | 8
  TOC | 17 | 7

15. Secondary Outcome: Proportion of Subjects in the m-MITT Populations With a With a Response of Overall Success (cUTI/AP)
Description: Proportion of subjects in m-MITT Population with response of cure and microbiological eradication or presumed eradication. Eradication defined for cUTI/AP as the demonstration that the bacterial pathogen(s) found at baseline is reduced to <10x4 CFU/mL urine (FDA). Clinical cure defined as complete resolution or significant improvement of the baseline signs & symptoms, no further antimicrobial warranted.
Time Frame: at EOT visit (7-14) and TOC visit (day 12-23)
Population: m-MITT Population (cUTI/AP Subjects Only)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 13 | 8
Participants
  EOT | 10 | 4
  TOC | 4 | 4

16. Secondary Outcome: Proportion of Subjects in the m-MITT Populations With a With a Response of Overall Success (Bacteremia Only)
Description: Proportion of subjects in m-MITT Population with response of cure and microbiological eradication or presumed eradication. Clinical cure defined as complete resolution or significant improvement of the baseline signs & symptoms, no further antimicrobial warranted.
Time Frame: at EOT visit (7-14) and TOC visit (day 12-23)
Population: m-MITT Population (Bacteremia Subjects Only)
Measure: Count of Participants; unit: Participants
Arm/Group | Vabomere | Best Available Therapy
Number analyzed (Participants) | 15 | 8
Participants
  EOT | 8 | 3
  TOC | 8 | 2

ADVERSE EVENTS:
Time Frame: Day 1 Through the Late Follow-Up Visit (LFU)- LFU defined as 14 days (+ or - 2 days) after the EOT Visit (7-14 days)
Arm/Group | Vabomere | Best Available Therapy
All-Cause Mortality (participants affected / at risk) | 10/50 | 6/25
Serious Adverse Events (participants affected / at risk) | 17/50 | 11/25
Other Adverse Events (participants affected / at risk) | 28/50 | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vabomere (N=50) | Best Available Therapy (N=25)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 2 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 2 | 0
Multi-organ Failure (General disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Enterococcal bacteremia (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Klebsiella Bacteremia (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 4
Septic Shock (Infections and infestations) | 1 | 4
Superinfection Bacterial (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Hemorrhage (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arterial Hemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Shock Hemorrhagic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vabomere (N=50) | Best Available Therapy (N=25)
Diarrhea (Gastrointestinal disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 4 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 1
Abdominal Distension (Gastrointestinal disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 2 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 5 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Sickle Cell Anemia with Crisis (Blood and lymphatic system disorders) | 0 | 1
Oral Candidiasis (Infections and infestations) | 2 | 1
Systemic Candida (Infections and infestations) | 3 | 0
Candiduria (Infections and infestations) | 1 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 1
Bacteremia (Infections and infestations) | 0 | 1
Perinephric Abscess (Infections and infestations) | 0 | 1
Pseudomonal Bacteremia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection Enterococcal (Infections and infestations) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 5 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin B Complex Deficiency (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 4 | 3
Hypertension (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 0 | 1
Extremity Necrosis (Vascular disorders) | 0 | 1
Asthenia (General disorders) | 0 | 2
Generalized Edema (General disorders) | 1 | 1
Hypothermia (General disorders) | 2 | 0
Infusion Site Phlebitis (General disorders) | 1 | 1
Edema Peripheral (General disorders) | 0 | 2
Pain (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 1
Transaminases Increased (Investigations) | 0 | 2
Urine Output Decreased (Investigations) | 2 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 1
Blood Fibrinogen Decreased (Investigations) | 0 | 1
Blood Urea Increased (Investigations) | 0 | 1
Electrocardiogram QT Prolonged (Investigations) | 0 | 1
Tremor (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1
Parasthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 3
Renal Impairment (Renal and urinary disorders) | 1 | 2
Hematuria (Renal and urinary disorders) | 1 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Extrasystoles (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Confusional State (Psychiatric disorders) | 0 | 2
Restlessness (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 1
Incision Site Pain (Injury, poisoning and procedural complications) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Penile Hemorrhage (Reproductive system and breast disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Enrollment Challenges required the Sponsor to terminate the study early which led to a smaller number of patients being enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-04-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT02168946/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT02168946/SAP_001.pdf